CLINICAL TRIAL: NCT04661293
Title: Expanded Access Program for Autologous Muscle Derived Cells (AMDCs)
Acronym: AMDC
Status: Available | Type: Expanded Access
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Other Study IDs: AMDC-EAP
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Autologous Muscle Derived Cells (AMDCs)

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to autologous muscle derived cells (AMDCs). Treating physicians may submit requests for expanded access to Cook MyoSite's investigational product by email to MYO-ExpandedAccess@CookMyoSite.com.

DETAILED DESCRIPTION:
Cook MyoSite, Inc. (Cook MyoSite) is committed to conducting rigorous, controlled clinical trials with variable inclusion and exclusion criteria based upon the indicated use under investigation. Participation in our clinical trials is the first and most preferable route to access our investigational product.

We understand that there may be patients with a serious, life-threatening disease or condition that have explored all other treatment options and are unable or ineligible to participate in our clinical trials. Expanded access, otherwise known as "compassionate use" or "pre-approval access," is a potential pathway to access an investigational product that a patient may otherwise be unable to receive.

Cook MyoSite will consider providing an investigational product to a qualified requesting physician currently licensed within the United States via the United States Food and Drug Administration's (FDA's) expanded access pathway outside of an active clinical trial when eligibility criteria are met.

ELIGIBILITY:
Eligibility Criteria:

1. The patient has a serious or life-threatening disease or condition with no satisfactory alternative.
2. Positive assessment that the anticipated benefits outweigh the risks to the patient.
3. Positive assessment that Cook MyoSite has an adequate supply of resources for producing the investigational product.
4. A determination that expanded access will not interfere with Cook MyoSite's ability to complete clinical trials in a timely fashion or which might otherwise delay marketing approval and ultimately availability to all patients.
5. The patient can undergo a muscle biopsy procedure(s).
6. The patient can undergo Cook MyoSite's required donor screening and testing.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Cook MyoSite, Inc., Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Cook MyoSite, Inc. Expanded Access Webpage — https://resources.cookmyosite.com/terms-and-conditions-of-sale-and-delivery-0
- See also: Cook MyoSite, Inc. Webpage — https://www.cookmyosite.com/